CLINICAL TRIAL: NCT01639274
Title: Prevalence of Chronic Obstructive Pulmonary Disease in HIV-patient Population
Brief Title: Human Immunodeficiency Virus (HIV)and Chronic Obstructive Pulmonary Disease (COPD)
Acronym: HIV and COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-PP-09
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COPD (Other)
  Interventions: Other: COPD prevalence

INTERVENTIONS:
Other: COPD prevalence — Determine prevalence of COPD

SUMMARY:
Highly active antiretroviral therapy (HAART) has considerably improved survival of HIV-infected patients. Opportunist diseases and cancers linked to immunodepression have largely regressed. Challenge is now the management of cardio-vascular diseases, nephrologic, neurologic, osteo-articular diseases, chronic hepatitis and cancer no linked to immunodepression. All this comorbidities are more reported in HIV-infected patients than in general non-HIV infected patients. Those are directly linked to the effect of chronic HIV-infection on ageing, metabolic effects of HAART, and way of life characterising this population.

Chronic obstructive pulmonary disease (COPD) results from tobacco consumption. Bronchial chronic infection, immunity, and ageing are also involved in the physiopathology of COPD. This disease has never been evaluated in a large prospective cohort of HIV-infected patients whereas there is a known increase of tobacco consumption and pulmonary infection in this population regardless to the general population.

Characterisation of COPD disease in HIV patients will allow us to make an hypothetic epidemiological link between HIV- HAART and COPD independently of tobacco consumption, and to study different physiopathologic hypothesis evocated in COPD genesis, like an accelerate pulmonary ageing.

DETAILED DESCRIPTION:
The management of HIV is mainly represented by its commorbidities (cardio-vascular disease, nephrologic, neurologic, osteo-articular disease, chronic hepatitis and cancer no linked to immunodepression). COPD prevalence has never been studied in HIV population. In consequence, there is no guideline about the screening, treatment or follow-up of COPD in HIV patients. However this population seems particularly at risk to develop COPD because of high tobacco consumption and accelerate ageing. Thus, we need an epidemiologic study to understand the prevalence of COPD in HIV population in order to organize a specific screening and follow-up. This is supported by an improvement of COPD if early managed. On top of that, COPD screening will increase awareness of HIV patients on the problematic of tobacco consumption.

ELIGIBILITY:
Inclusion criteria:

* HIV seropositivity
* Age > 18 years
* Written aggreeing
* Affiliated or profit of a social coverage

Non inclusion criteria:

* Age < 18 years old
* Actual infectious pneumonia
* COPD exacerbation last 2 months *
* Recent (less than 1 month) myocardial infarction
* Thoracic or abdominal pain
* Enable to answer question secondary to mental deficienty**
* Physic or mental incapacity to realise COPD-6 or spirometery
* Urinary incontinency with effort
* Prisoner
* Refuse of consent or incapacity to give his consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of Chronic obstructive pulmonary disease prevalence in a large population of HIV patients | one time each patient (one hour)
  An auto-questionnaire will be given to each patient included in the study (concern respiratory symptoms, tobacco consummation, illicit drug use, various respiratory exposition and lifestyle). Each patient will release a rapid evaluation of respiratory capacity with COPD-6. Patients screened with abnormal respiratory symptoms on auto-questionnaire, or with a risk of COPD ranked from high to moderate by COPD-6 test will benefit of a conventional spirometry.

SECONDARY OUTCOMES:
Epidemiological characteristics of COPD in HIV population | one time each patient (1 hour)
  Epidemiological characteristics of COPD in HIV population: age, severity of the disease compared to the GOLD classification, symptoms of chronic bronchitis, exacerbation frequency, immune statute, HAART exposure, lung opportunist infection, tobacco consumption, cannabis and others drugs consumption, professional exposition..Descriptive comparison of respiratory risk factors, immunity and HAART exposition between HIV patients with and without COPD.Define proportion of under-diagnose COPD in HIV population.

CONTACTS AND LOCATIONS:
Overall Officials: Karine RISSO, MD, Principal Investigator — CHU NICE
Locations (1):
- Service d'Infectiologie - Hôpital de l'Archet, Nice, France